CLINICAL TRIAL: NCT04567485
Title: Impact of Moderate to Severe Pain in the Post-intervention Monitoring Room After Hemorrhoidectomy on the Length of Stay in the Outpatient Surgery Unit
Acronym: HEM_DOULEUR
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: HEM_DOULEUR
Record Dates: First submitted 2020-09-17; First posted 2020-09-28 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Hemorrhoids; Surgery
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The target rate for outpatient surgery has been set by the Ministry of Health at 70% for 2020. To achieve this objective, this requires increasing the panel of eligible outpatient procedures to more mutilating surgeries and usually performed in conventional hospitalization. This switch from conventional hospitalization to an outpatient stay increases the risk of converting stays into unscheduled hospitalization. Postoperative pain is one of the main factors in converting outpatient stays. Poor control is associated with increased length of stay, and unscheduled consultations and readmissions. In addition, the increased time spent with severe pain during the first 24 hours postoperatively is a risk factor for chronicization.

Proctology, and, in particular, hemorrhoidal surgery is the perfect example. Outpatient management of open pedicle hemorrhoidectomy is increasing year by year, but the rate of conversion to unscheduled hospitalizations remains high. Urine retention, postoperative hemorrhage and poor pain control are the main causes. Within the Paris Saint Joseph Hospital Group, hemorrhoidal surgery has the highest rate of conversions from hospitalization to proctology (8% in 2019), despite the implementation since 2015 of a dedicated, developed according to the current recommendations of the SNFCP.

The pain after hemorrhoidal surgery is always severe in the absence of analgesics and appears upon arrival in the post-interventional monitoring room (SSPI). Despite the administration of analgesics or the implementation of locoregional analgesia techniques (pudendal block), moderate to severe pain is frequently observed in the post-intervention monitoring room. In the medical literature, there is little data evaluating the means of management of postoperative pain in this surgery, and even less the effect of the different associations.

Retrospectively and, from the data collected in our information systems, we wish to assess the impact on the length of stay of the presence of moderate to severe pain in the IPSS after a two-way or tri-pedicle hemorrhoidal surgery open on our cohort of patients operated in outpatient surgery. Our hypothesis is that the presence of moderate to severe pain in PPSS increases the total length of stay, placing the patient at an increased risk of conversion. The purpose of our study is also to identify predictive factors (aggravating or protective) of the onset of moderate to severe pain immediately after surgery, in order to establish a strategy to limit its frequency.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age is ≥ 18 years
* Patient scheduled for outpatient hospitalization,
* Patient operated on for open hemorrhoidectomy surgery, between January 01, 2019 and December 31, 2019
* French-speaking patient

Exclusion Criteria:

* Patient scheduled for conventional hospitalization
* Patient not having an anesthesia report in DxCare®
* Patient not having a report of passage in SSPI in DxCare ®
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under legal protection
* Patient objecting to the use of his medical data in the context of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be carried out on data from patients operated on for open outpatient hemorrhoidectomy surgery within the Groupe Hospitalier Paris Saint-Joseph, between January 01, 2019 and December 31, 2019, i.e. 450 patients in total.
Sampling Method: Non-Probability Sample
Enrollment: 446 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Impact of moderate to severe pain postoperatively from an open bi- or tri-pedicular hemorrhoidectomy scheduled on an outpatient basis | Day 30
  This outcome corresponds to the total length of stay of the patient within the Paris Saint Joseph Hospital, obtained by calculating the difference between the date and time of discharge from the hospital, and the date and time of entry into the Ambulatory Surgery Unit .

SECONDARY OUTCOMES:
Length of stay in SSPI | Day 30
  This outcome corresponds to the duration of stay in SSPI calculated from the difference between the time of exit and the time of entry into SSPI.
Conversion rate from hospital to outpatient to conventional hospitalization | Day 30
  This outcome corresponds to the conversion rate calculated by the ratio between the number of patients whose scheduled outpatient stay is transformed into conventional hospitalization over the total number of patients scheduled as outpatient.
Independent predictive factors that reduce or increase the risk of moderate to severe pain | Day 30
  This outcome corresponds to the evaluatiob of predictive factors that reduce or increase the risk of moderate to severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal ALFONSI, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Result] American Society of Anesthesiologists Task Force on Acute Pain Management. Practice guidelines for acute pain management in the perioperative setting: an updated report by the American Society of Anesthesiologists Task Force on Acute Pain Management. Anesthesiology. 2012 Feb;116(2):248-73. doi: 10.1097/ALN.0b013e31823c1030. No abstract available. PMID 22227789
- [Result] Vinson Bonnet B, Juguet F; French National Coloproctology Society. Ambulatory proctologic surgery: Recommendations of the French National Coloproctology Society (SNFCP). J Visc Surg. 2015 Dec;152(6):369-72. doi: 10.1016/j.jviscsurg.2015.10.001. Epub 2015 Nov 5. No abstract available. PMID 26547481
- [Result] Joshi GP, Neugebauer EA; PROSPECT Collaboration. Evidence-based management of pain after haemorrhoidectomy surgery. Br J Surg. 2010 Aug;97(8):1155-68. doi: 10.1002/bjs.7161. PMID 20593430
- [Result] Sammour T, Barazanchi AW, Hill AG; PROSPECT group (Collaborators). Evidence-Based Management of Pain After Excisional Haemorrhoidectomy Surgery: A PROSPECT Review Update. World J Surg. 2017 Feb;41(2):603-614. doi: 10.1007/s00268-016-3737-1. PMID 27766395